CLINICAL TRIAL: NCT04429724
Title: Health Professional Exposure Assessment to Covid-19
Acronym: SERODRON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RIPH_2020_8
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- health workers at hospital (Experimental): Three blood samples will be taken at day 1, month 3 and month 6. A prospective data collection will be set up at the level of symptoms and co-morbidities at each collection at D1, M3 and M6.
  Interventions: Diagnostic Test: Diagnostic test Covid-19

INTERVENTIONS:
Diagnostic Test: Diagnostic test Covid-19 — Three blood samples will be taken at day 1, month 3 and month 6 A prospective data collection will be set up at the level of symptoms and co-morbidities at each collection at D1, M3 and M6.

SUMMARY:
Understanding the SARS-Cov2 epidemic is a major public health issue, both in the community and in the hospital sector. Because of their central position in the management of patients infected with COVID-19, hospital staff may be considered at high risk of infection. The development of serological tests makes it possible to reliably document a contamination, symptomatic or not, that is more than 3 weeks old. These tests, combined with clinical questioning of the symptoms, make it possible to determine the proportion of asymptomatic infections whose impact in the transmission of this disease appears to be major. The duration of the presence of the antibodies that are hoped to neutralize after infection with CoV2-SARS remains uncertain. Documenting the evolution of antibody levels and their monitoring in a population at high risk of re-exposure to CoV2-SARS is a major issue in understanding this disease and in assessing the risk of infection among healthcare workers.

DETAILED DESCRIPTION:
This is a multi-center, prospective, interventional, low-risk, low-constraint, biological collection study to assess the exposure of health care workers to COVID-19.

Three blood samples will be taken at day 1, month 3 and month 6. The blood samples will be stored in a serum biological collection. A prospective data collection will be set up at the level of symptoms and co-morbidities at each collection at D1, M3 and M6.

In the event of the appearance of symptoms between samples, a self-questionnaire will be completed by the participating personnel as well as an invitation to screening by RT-PCR SARS Cov2 according to standard practices in force at the national level as well as an additional serological test.

ELIGIBILITY:
Inclusion Criteria:

* Staff on duty in the health facility
* Eligible to be drawn
* Beneficiary subject affiliated or entitled to a social security scheme

Exclusion Criteria:

* Minor patient
* Refusal to participate
* Patient under guardianship
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2129 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Number of contaminated personnel | day 1
  Number of contaminated personnel by occupational category and department on day 1.

SECONDARY OUTCOMES:
Number of contaminated personnel | month 3
  Number of contaminated personnel by professional category and by service at month 3 a by serological test
Number of contaminated personnel | month 6
  Number of contaminated personnel by professional category and by service at month 6 a by serological test
Number of symptomatic staff by occupational category and service | month 3
  Number of symptomatic staff by occupational category and service at Month 3 with positive RT-PCR Cov2 SARS
Number of symptomatic staff by occupational category and service | month 6
  Number of symptomatic staff by occupational category and service at Month 6 with positive RT-PCR Cov2 SARS
Number of contaminated personnel with effective protection | evolution at day 1, month 3 and month 6
  Number of contaminated personnel with effective protection: evolution of the antibody index at day 1, month 3 and month 6
comparison of socio-demographic characteristics and co-morbidities between patients losing their antibodies and those maintaining their antibodies | month 6
  comparison of socio-demographic characteristics and co-morbidities between patients losing their antibodies and those maintaining their antibodies between two stitch dates.

CONTACTS AND LOCATIONS:
Overall Officials: PATOZ Pierre, PharmD, Principal Investigator — CH TOURCOING
Locations (4):
- France (4):
  - CH Roubaix, Roubaix
  - CH Tourcoing, Tourcoing
  - CH Wasquehal, Wasquehal
  - CH Wattrelos, Wattrelos

IPD SHARING:
Plan to Share IPD: No